CLINICAL TRIAL: NCT06079099
Title: Time Within the Acute Care Chain: How Long Have Medical Emergency Department Patients Spent
Acronym: TACC
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: TACC
Record Dates: First submitted 2021-12-22; First posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2021-12

CONDITIONS: Emergencies
Keywords: Acute Care Chain; Emergency Department; Patient Journey
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is part of a research domain focusing on the acute care chain, which includes the patient journey from symptoms to treatment on the Emergency Medical Department (ED). Within hospitals there is much attention for triage and the amount of time patients spent within the chain, especially for the ED. However, there is less information available on what occurs before patients visit the ED. Gaining more insight in the patient journey in the acute care chain as a whole, might provide important information to further optimize care at the ED. In the current study, 750 patients will be included at multiple ED's in the Netherlands. The primary goal is to gain insight in the patient journey of adult ED patients.

DETAILED DESCRIPTION:
All adult ED patients in the province of Limburg will be included in a 72 hour time frame. Students were present at the EDs 24 hours to include all these patients. Patient data were gathered from medical records (including hospital file, referral letters and EMS notes) using a Case Report Form (CRF) and from a questionnaire filled out by the patient. Data were collected on demographic variables, including sex, age, highest level of education, living situation and the presence of roommates. Furthermore, information regarding the ACC and Time spent in the ACC (TACC) was collected.

The entire ACC was divided into four phases: the pre-referral phase, the referral phase, the ED phase and the post ED phase. In each phase several variables were collected.

Pre-referral phase The pre-referral phase started with the onset of complaints this disease period up to the referring contact. The following variables of this phase were collected: the symptom duration in days calculated from the day of onset of symptoms until ED visit, number of prior contacts with a healthcare provider and prescribed medication this disease period before ED visit. A prior contact with a healthcare provider was defined as a contact within this disease period, regarding the same complaint, and before the contact during which the patient was referred to the ED.

Referral phase The referral phase started with the moment of referral until arrival at the ED. The following variables of this phase were collected: time and date of referral contact, referring health care provider (GP, EMS, medical specialist, nursing home doctor, other or self-referral), prehospital triage urgency (EMS and GCP), and mode of transportation to the ED (own transport or by EMS). Prehospital triage urgency levels (for GPC and EMS) are determined using the Netherlands Triage Standard (NTS), which categorizes patients from U1 (life threatening, immediate action required) up to U5 (advice, a physical examination can wait until the next day) (16). If necessary, an ambulance is subsequently dispatched according to these urgency levels.

ED phase The ED phase started with arrival at the ED until hospital discharge, including 30-day follow-up. The following variables of this phase were collected at the ED: referred specialty (the specialty to which the patient has been referred), treating specialty (the specialty that eventually treated/discharged/admitted the patient), triage urgency level (MTS (17)), presenting symptoms, the number of patients with a presumptive prespecified complex condition, ED work up, and arrival and departure time in the ED to calculate the length of stay (LOS).

The EDs in this study use the Manchester Triage System (MTS) as a triage system, which categorises patients into five levels of urgency (17). Immediate (red) patients are to be evaluated immediately, whereas non-urgent (blue) patients are allowed to wait for 240 minutes prior to evaluation. In this study we combined red and orange triage urgencies as 'highly urgent' (evaluation within 10 minutes maximum), and yellow, green and blue as 'urgent' (evaluation within 60-240 minutes). Presenting symptoms were categorized into 18 groups after discussion with the researchers: minor trauma, abdominal pain, dyspnoea, general malaise, fever, extremity complaints (e.g. arthritis), neurological complaints, syncope/palpitations, skin symptoms, urological complaints, complaints after treatment, allergic reaction, hypertension, minor oncological complaints (e.g. rash), chest pain, ENT problem, intoxication, and other. Prespecified complex conditions were defined as patients presenting with the presumptive diagnosis of a stroke, myocardial infarction, aortic syndrome or major trauma.

The ED work up was defined as simple when ED work-up included lab tests, electrocardiogram and X-ray and was defined complex when included CT, ultrasound, lumbar puncture (LP), abdominal paracentesis, gastroscopy, MRI scan and consultations of other specialties.

Post ED phase The post ED phase started after ED discharge until 30-day follow-up. The following variables were collected: post-ED disposition, 7- and 30-day all-cause mortality and 30-day revisit. A combination of 7- and 30-day all-cause mortality and 30-day revisit were called adverse outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients of 18 years and older
* Patient is treated at ED during inclusion period
* Patient is able and willing to sign informed consent or has a legal representative

Exclusion Criteria:

- Language barrier

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients who visit the ED in need of acute care
Sampling Method: Probability Sample
Enrollment: 583 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2022-04-24 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Total time a patient spent in acute care chain. | up to hours with a maximum of 48 hours.Time unit: hours.
  Patient journey in the acute care chain. From all included patients: We measure the duration in the Acute care chain: From the moment a patient has contact with the referring healthcare provider until ED discharge

SECONDARY OUTCOMES:
Number of contacts with a healthcare provider this disease period | Days, maximum 14 days. Time unit: days.
  Did patients have contact with care provider(s) before visiting the ED? If yes, which type of care providers were they and what was the urgency level? We ask the included patients during the inclusion periode how many healthcare providers the contacted: From first contact with a healthcare provider this disease period until entering the ED. This disease period = start complaints
How many investigations were done during the ED visit | During ED stay, that means in a couple of hours. ED stays are no longer that > 1 day. time unit is hours.
  Which investigations are carried out: blood test, ultrasound, x-ray? Patients that present in the inclusion period, at the ED. During the ED visit of the patient we look at the amount and which ancillary investigations are done. Timeframe = ED stay. No change is measured.
Number of participant that are admitted to the hospital. | 30 days after ED visit we check on how many patients are admitted. Time frame 30 days. Unit: number of participants.
  What happens after ED visit? How many patients will be admitted.
Number of participant that are deceased after 30 days. . | 30 days after ED visit we check on how many patients are deceased. Time frame 30 days. Unit: number of participants.
  What happens after ED visit? How many patients died

CONTACTS AND LOCATIONS:
Locations (6):
- Netherlands (6):
  - MUMC, Maastricht, Limburg
  - Zuyderland MC, Heerlen
  - Laurentius Ziekenhuis Roermond, Roermond
  - Zuyderland MC, Sittard
  - VieCuri, Venlo
  - St. Jans Gasthuis Weert, Weert

REFERENCES:
- [Derived] Claassen L, Stassen PM, Boumans TJT, Barten DG, Kremers MNT, Hermans AME, Zelis N, Cals JWL, Latten GHP. Characteristics of Dutch ED patients and their journey through the acute care chain: A province-wide flash-mob study. PLoS One. 2025 Apr 3;20(4):e0318510. doi: 10.1371/journal.pone.0318510. eCollection 2025. PMID 40179077

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-17): https://cdn.clinicaltrials.gov/large-docs/99/NCT06079099/Prot_SAP_000.pdf
  • Informed Consent Form (2021-08-13): https://cdn.clinicaltrials.gov/large-docs/99/NCT06079099/ICF_001.pdf